CLINICAL TRIAL: NCT07272499
Title: A Prospective, Multicenter, Open-Label Clinical Study of Orelabrutinib Plus Lisaftoclax and Rituximab in Treatment-Naive, High-Risk Mantle Cell Lymphoma (MCL)
Brief Title: Orelabrutinib Plus Lisaftoclax and Rituximab in Untreated Mantle Cell Lymphoma With High-Risk Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Fujian Medical University Union Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Third Xiangya Hospital of Central South University (Other); Qilu Hospital of Shandong University (Other); Shanghai Minhang Central Hospital (Other); Huadong Hospital (Other); Yangpu District Central Hospital Affiliated to Tongji University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Order2-HR
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-09

CONDITIONS: Mantle Cell Lymphoma (MCL)
Keywords: Order2
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — orelabrutinib; Rituximab; Lisaftoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib + Lisaftoclax + Rituximab and Orelabrutinib + Lisaftoclax Maintenance (Experimental): 1. In induction phase, patients will receive rituximab 375 mg/m² IV on day 1/cycle; orelabrutinib 150 mg/day PO once daily; and lisaftoclax PO Cycle1(100mg day1, 200mg day2, 400mg day3, 600mg/day day4-28), Cycle2-6 600mg/day, every 28 day per cycle for 6 cycles.
  2. In maintenance phase, Patients with an objective response (complete or partial) after induction therapy will recieve orelabrutinib 150 mg/day PO once daily and lisaftoclax 600mg/day PO once daily, every 28 day per cycle for 24 cycles.
  Interventions: Drug: Orelabrutinib; Drug: Rituximab (R); Drug: Lisaftoclax (APG-2575)

INTERVENTIONS:
Drug: Orelabrutinib — 150mg/day PO once daily
  Other Names: Induction phase
Drug: Rituximab (R) — 375 mg/m² IV on day 1/cycle
  Other Names: Induction phase
Drug: Lisaftoclax (APG-2575) — Cycle1(100mg day1, 200mg day2, 400mg day3, 600mg/day day4-28), Cycle2-6 600mg/day, PO once daily.
  Other Names: Induction phase
Drug: Lisaftoclax (APG-2575) — 600mg/day, PO once daily
  Other Names: Maintenance phase

SUMMARY:
This multicenter, open-label, trial aims to evaluate the efficacy and safety of orelabrutinib plus lisaftoclax and rituximab in patients with high-risk mantle cell lymphoma (MCL). The primary objective is to assess the optimal complete response (CR) rate during the induction phase, with secondary objectives including progression-free survival (PFS), overall survival (OS), objective response rate (ORR), and safety. Exploratory analysis will investigate the correlation between tumor biomarkers and treatment efficacy.

DETAILED DESCRIPTION:
Mantle cell lymphoma (MCL) is an aggressive B-cell malignancy accounting for 2-10% of non-Hodgkin lymphomas, primarily affecting middle-aged and elderly individuals. Conventional immunochemotherapy often yields suboptimal outcomes in high-risk subtypes, such as those with blastoid variant morphology, high MIPI score, Ki-67 >30%, TP53 abnormalities, or complex karyotype . Over the past decade, the approval of targeted agents has introduced novel combination regimens, offering new therapeutic avenues for these patients.

The SYMPATICO trial demonstrated that ibrutinib combined with venetoclax significantly prolonged progression-free survival (PFS) in patients with relapsed/refractory (R/R) MCL compared to placebo after a median follow-up of 51.2 months. Subgroup analysis revealed a pronounced benefit in TP53-mutated patients (HR 0.57, 95% CI 0.33-0.97). Among 74 TP53-mutated patients receiving the combination, median PFS was 20.9 months, with a complete response (CR) rate of 57% and a duration of CR of 32.2 months. The BoVen regimen (BTK inhibitor + obinutuzumab + venetoclax) reported a CR rate of 88% in 25 treatment-naïve TP53-mutated MCL patients. After a median follow-up of 28.2 months, the 2-year PFS rate was 72%, outperforming outcomes in the SYMPATICO TP53-mutant cohort. These results underscore the promise of combining BTK inhibitor, anti-CD20 antibody, and Bcl-2 inhibitor, not only for TP53-mutant high-risk groups but potentially for a broader patient population.

Lisaftoclax is a next-generation Bcl-2 inhibitor with efficacy comparable to venetoclax but featuring an improved safety profile and more convenient dosing. It has been approved in China and is currently in international Phase III trials for CLL/SLL, MDS, and AML. Orelabrutinib is a novel, highly selective BTK inhibitor associated with reduced off-target effects and enhanced safety. Large-scale, non-head-to-head safety comparisons suggest it has a favorable safety standing in its class. Therefore, this study is planned to evaluate the efficacy and safety of orelabrutinib in combination with lisaftoclax and rituximab for high-risk MCL. High-risk factors include blastoid/pleomorphic variant, TP53 mutation/loss or p53 protein expression >50%, Ki-67 ≥30%, and high-risk MIPI status.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MCL (mantle cell lymphoma) through flow cytometry or histopathology, and has not received prior treatment.
* Age > 14 years of age, both genders are eligible.
* Ann Arbor stage II-IV; for stage II subjects, those who require systemic therapy based on the investigator's judgment are eligible.
* At least one measurable lesion.
* Any one of the following high-risk factors is present: MIPI score of 6-11, Ki67 > 30%, TP53 mutation/loss or p53 protein expression >50%, blastic or pleomorphic variation.
* Laboratory tests (blood routine, liver and kidney function) meet the following requirements: a) Blood routine: White blood cell count ≥3.0×10^9/L, absolute neutrophil count ≥1.5×10^9/L, hemoglobin ≥90g/L, platelet count ≥75×10^9/L. b) Liver function: Transaminases ≤2.5 times the upper limit of normal, bilirubin ≤1.5 times the upper limit of normal. c) Serum creatinine 44-133 mmol/L.
* The investigator judges that the subject's life expectancy is greater than 12 weeks from the time of screening.
* Willing and able to participate in all required assessments and procedures of the study protocol.

Exclusion Criteria:

* Patients who have previously received treatment with BTK inhibitors.
* Patients with severe complications or serious infections.
* Patients with uncontrolled cardiovascular diseases, coagulation disorders, connective tissue diseases, serious infectious diseases, etc.
* Patients with active infections requiring systemic treatment, including bacterial, fungal, and viral infections.
* HIV-infected individuals.
* Patients with mental disorders or those who are known or suspected to be unable to fully comply with the study protocol.
* Patients whom the investigator judges to have other conditions that make them unsuitable for participation in this study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2028-09-10 (Estimated); Study Completion 2028-09-10 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | End of induction treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=28 days]
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Overall Response Rate | End of induction treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=28 days]
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Progression-free survival | Baseline up to data cut-off (up to approximately 3 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off (up to approximately 3 years)
  Overall survival was defined as the time from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No